CLINICAL TRIAL: NCT05774509
Title: Treatment of Non-ischemic Dilated Cardiomyopathies by Intravenous Infusions of the Extracellular Vesicle-Enriched Secretome of Cardiovascular Progenitor Cells
Brief Title: Treatment of Non-ischemic Cardiomyopathies by Intravenous Extracellular Vesicles of Cardiovascular Progenitor Cells
Acronym: SECRET-HF
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APHP200034; 2022-001844-75 (EudraCT Number); PHRC-19-0330 (Other Grant/Funding Number: French ministry of health)
Record Dates: First submitted 2023-02-20; First posted 2023-03-17 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Heart Failure With Reduced Ejection Fraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treated group (Experimental): A maximum of 12 patients will be included in the study following a dose-escalating design:
  * Cohort 1 (4 patients) will receive 20x10E9 particles/kg for each infusion, with a total of 3 infusions, for a cumulative dose of 60x10E9 particles/kg;
  * Cohort 2: in the absence of safety issues in Cohort 1, 8 patients will receive 40x10E9 particles/kg for each infusion, with a total of 3 infusions, for a cumulative dose of 120x10E9 particles/kg.
  Interventions: Biological: Extracellular vesicle-enriched secretome of cardiovascular progenitor cells differentiated from induced pluripotent stem cells

INTERVENTIONS:
Biological: Extracellular vesicle-enriched secretome of cardiovascular progenitor cells differentiated from induced pluripotent stem cells — Repeated (X3) intravenous infusions of the extracellular vesicle-enriched secretome of cardiovascular progenitor cells (differentiated from human induced pluripotent stem cells)

SUMMARY:
The goal of this clinical trial is to assess the safety and efficacy of three intravenous injections of the extracellulat vesicle-enriched secretome of cardiovascular progenitor cells in severely symptomatic patients with drug-refractory left ventricular (LV) dysfunction secondary to non-ischemic dilated cardiomyopathy. The main questions it aims to answer are:

* Are these repeated injections safe and well tolerated?
* Do they improve cardiac function and, if yes, to what extent?

DETAILED DESCRIPTION:
The overall objective of this study is to assess the safety and efficacy of repeated intravenous injections of the secretome of cardiovascular progenitor cells in severely symptomatic patients with drug-refractory left ventricular (LV) dysfunction secondary to non-ischemic dilated cardiomyopathy.

The rationale and design of this trial are based on three main assumptions:

1. The tissue-repair capacity of transplanted cells can be duplicated by the delivery of the extracellular vesicles (EV) that they secrete.
2. The greatest therapeutic efficacy seems to be achieved by using secreting cells that are committed to the same lineage as those of the tissue to be repaired, hence, the use of cardiovascular progenitor cells as the source of the EV-enriched secretome.
3. Leveraging the benefits of cells, or their secreted products, by repeated administrations requires a non-invasive approach, which highlights the potential interest of the intravenous approach.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 to 80 years
2. Signed written informed consent
3. French Social Security affiliation;
4. Dilated cardiomyopathy defined by a dilated LV with a reduced EF ≤40% on echocardiography and/or CMR imaging, unexplained by pressure or volume overload (severe arterial hypertension or significant valve disease), coronary artery disease (as assessed by coronary angiography) or a systemic disease; in case of chemotherapy-induced cardiomyopathy, patients should have a period of at least two years of clinical cancer-free state* and a low estimated likelihood of recurrence (≤30% at 5 years), as determined by an oncologist, based on tumor type, response to therapy, and negative metastatic work-up at the time of diagnosis (*exceptions to this are carcinoma in situ or fully resected basal and squamous cell cancer of the skin);
5. NYHA Class III in spite of optimal heart failure maximally tolerated guideline-directed medical therapy, including cardiac resynchronization if needed, without other treatment options;
6. Plasma level of B-type natriuretic peptide (BNP) > 150 pg/mL or, N-terminal pro-BNP (NT-proBNP) ≥ 400 pg/mL;
7. For child-bearing aged women, efficient contraception such as combined (estrogen and progestogen containing) hormonal contraception or progestogen-only hormonal contraception associated with inhibition of ovulation and for men efficient contraception such as condom, during treatment and until the end of the relevant systemic exposure, i.e. until 3 months after the end of treatment.

Exclusion Criteria:

1. Implantation of a cardiac resynchronisation therapy device or an ICD unit during the preceding 3 months;
2. End-stage heart failure with reduced EF (HFrEF) defined as patients with American College of Cardiology Foundation/American Heart Association (ACCF/AHA) stage D (candidates for specialized interventions, including heart transplantation and mechanical assistance) or terminal HF (advanced HF with poor response to all forms of treatment, frequent hospitalizations and life expectancy < 12 months)
3. Patients treated with inotropic agents during the 1 month period prior to inclusion;
4. Acute heart failure (regardless of the cause);
5. Heart failure caused by cardiac valve disease, untreated hypertension or documented coronary artery disease with lesions which could explain the cardiomyopathy;
6. Cardiomyopathy due to a reversible cause e.g. endocrine disease, alcohol or drug abuse, myocarditis, Tako-Tsubo, or arrhythmias;
7. Cardiomyopathy due a syndromic/systemic disease (e.g. Duchenne's muscular dystrophy, immune/inflammatory/infiltrative disorders [amyloidosis, hemochromatosis]);
8. If post-chemotherapy cardiomyopathy: a history of radiation therapy AND evidence of constrictive physiology; a baseline computerized tomography scan or CMR showing new tumor or suspicious lymphadenopathy raising concern of malignancy; a trastuzumab treatment within the last 3 months;
9. Previous cardiac surgery;
10. Recent stroke (within the last 3 months);
11. Documented presence of a known LV thrombus, aortic dissection, or aortic aneurysm;
12. Uncontrolled ventricular tachycardia defined by sustained ventricular tachycardia, including electrical storm and incessant ventricular tachycardia with no response to antiarrhythmic medication; Internal Cardioverter Defibrillator firing in the 30 days prior to the first infusion;
13. History of drug-induced allergic reactions or allergy of any type having required treatment;
14. Contraindication to corticosteroids or anti-histaminic agents;
15. Contraindication to gadoterate meglumine if it will be used with CMR;
16. Hematological disease: anaemia (haematocrit < 25%), leukopenia (leucocytes < 2,500/μL) or thrombocytopenia (thrombocytes < 100,000/μL); myeloproliferative disorders, myelodysplastic syndrome, acute or chronic leukaemia, and plasma cell dyscrasias (multiple myeloma);
17. Coagulopathy not due to a reversible cause;
18. Diminished functional capacity for other reasons such as: Chronic Obstructive Pulmonary Disease (COPD) with Forced Expiratory Volume (FEV) <1 L/min, moderate to severe claudication or morbid obesity;
19. Diabetes with poorly controlled blood glucose levels and/or evidence of proliferative retinopathy;
20. Dialysis-dependent renal insufficiency;
21. Autoimmune disorders or current immunosuppressive therapy;
22. History of organ transplant or cell-based treatment;
23. Serum positivity for HIV, hepatitis BsAg, or viremic hepatitis C;
24. Female patient who is pregnant, nursing, or of child-bearing potential and not using effective birth control;
25. Active infection;
26. Known allergy to aminoglycosides;
27. Patient under legal protection (guardianship);
28. Participation in another interventional trial;
29. Life expectancy less than one year.
30. Contraindication to 18FDG-PETscan

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-05-31 (Actual); Primary Completion 2025-08-15 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Serious Adverse Events | 10 weeks after the onset of treatment: 6 weeks of treatment and 4 weeks of follow-up after the last IMP infusion.
  Number of any potentially Serious Adverse Events (SAEs)/Reactions attributed to the experimental treatment: death (cardiovascular or of any cause), hospitalization for worsening heart failure, acute coronary syndrome (including myocardial infarction), sustained atrial and ventricular arrhythmias, ischemic stroke, immune-allergic or infectious reactions to the intravenous infusions of the IMP, and any other potential adverse effects detected and corroborated by clinical presentation, laboratory investigations and image analysis.

SECONDARY OUTCOMES:
Validation of the bioactivity of the EV-enriched secretome by proliferation of human vascular endothelial cells. | 12 months
  Bioactivity of the IMP (potency tests) assessed by proliferation of human vascular endothelial cells assessed by BrdU (>20% relative to the control).
Validation of the bioactivity of the EV-enriched secretome by activation of allogeneic peripheral blood mononuclear cells. | 12 months
  Bioactivity of the IMP (potency tests) assessed by activation of allogeneic peripheral blood mononuclear cells assessed by the secretion of IL-2 and IFNγ (lack of increased secretion compared with the control).
Validation of the bioactivity of the EV-enriched secretome | 12 months
  Bioactivity of the IMP (potency tests) assessed by degranulation of Natural Killer cells assessed by the expression of CD107 (compared with a negative control).
Assessment of the effects of the IMP on immune and inflammatory responses at 3 weeks after the onset of the treatment. | 3 weeks after the onset of the treatment.
  Detection of donor-specific antibodies before the second secretome infusion.
Assessment of the effects of the IMP on immune and inflammatory responses at 6 weeks after the onset of the treatment. | 6 weeks after the onset of the treatment.
  Detection of donor-specific antibodies before the third secretome infusion.
Assessment of the effects of the IMP on immune and inflammatory responses at 10 weeks after the onset of the treatment. | 10 weeks after the onset of the treatment.
  Detection of donor-specific antibodies at 28 days following the last secretome infusion.
Assessment of the effects of the IMP on immune and inflammatory responses at 6 months after the last secretome infusion. | 6 months after the last secretome infusion.
  Detection of donor-specific antibodies at 6 months following the last secretome infusion if DSA are detected at the 28 days post-treatment study point at MFI ≥ 5000.
Inflammatory response to IMP infusions | 28 days, 6 and 12 months following the third infusion
  Assessment of blood levels of interleukins, C- Reactive Protein and immune cells.
Monitoring for Major Cardiovascular Adverse Events (MACE) | 28 days following the last IMP infusion and subsequently until 1 year after the end of treatment
  MACE including cardiac death, rehospitalization for heart failure, acute coronary syndromes, ischemic stroke and ventricular arrhythmias during the 1-year follow-up.
Changes in LV function assessed by NYHA at 28 days after the end of the treatment. | 28 days after the end of the treatment.
  New York Heart Association (NYHA) functional class.
Changes in LV function assessed by NYHA at 6 months after the end of the treatment. | 6 months after the end of the treatment.
  New York Heart Association (NYHA) functional class.
Changes in LV function assessed by NYHA at 12 months after the end of the treatment. | 12 months after the end of the treatment.
  New York Heart Association (NYHA) functional class.
Changes in LV function assessed by Minnesota Living With Heart Failure questionnaire at 6 months after the end of the treatment. | 6 months after the end of the treatment.
  Quality of life assessed by Minnesota Living With Heart Failure questionnaire.
Changes in LV function assessed by Minnesota Living With Heart Failure questionnaire at 12 months after the end of the treatment. | 12 months after the end of the treatment.
  Quality of life assessed by Minnesota Living With Heart Failure questionnaire.
Changes in LV function assessed by LV ejection fraction at 28 days after the end of the treatment. | 28 days after the end of the treatment.
  Measurements of LV ejection fraction (EF%) by Doppler-echocardiography.
Changes in LV function assessed by LV ejection fraction at 6 months after the end of the treatment. | 6 months after the end of the treatment.
  Measurements of LV ejection fraction (EF%) by Doppler-echocardiography.
Changes in LV function assessed by LV ejection fraction at 12 months after the end of the treatment. | 12 months after the end of the treatment.
  Measurements of LV ejection fraction (EF%) by Doppler-echocardiography.
Changes in LV function assessed by LV Volumes at 28 days after the end of the treatment. | 28 days after the end of the treatment.
  LV Volumes ml/m2 by Doppler-echocardiography.
Changes in LV function assessed by LV Volumes at 6 months after the end of the treatment. | 6 months after the end of the treatment.
  LV Volumes ml/m2 by Doppler-echocardiography.
Changes in LV function assessed by LV Volumes at 12 months after the end of the treatment. | 12 months after the end of the treatment.
  LV Volumes ml/m2 by Doppler-echocardiography.
Changes in LV function assessed by LV global longitudinal strain at 28 days after the end of the treatment. | 28 days after the end of the treatment.
  LV global longitudinal strain (%) by Doppler-echocardiography.
Changes in LV function assessed by LV global longitudinal strain at 6 months after the end of the treatment. | 6 months after the end of the treatment.
  LV global longitudinal strain (%) by Doppler-echocardiography.
Changes in LV function assessed by LV global longitudinal strain at 12 months after the end of the treatment. | 12 months after the end of the treatment.
  LV global longitudinal strain (%) by Doppler-echocardiography.
Changes in LV function assessed by LV ejection fraction (%) by Cardiac Magnetic Resonance at 6 months after the end of the treatment. | 6 months after the end of the treatment.
  Measurements of LV ejection fraction (%) by Cardiac Magnetic Resonance.
Changes in LV function assessed by LV ejection fraction (%) by Cardiac Magnetic Resonance at 12 months after the end of the treatment. | 12 months after the end of the treatment.
  Measurements of LV ejection fraction (%) by Cardiac Magnetic Resonance.
Changes in LV function assessed by LV volumes (ml/m2) by Cardiac Magnetic Resonance at 6 months after the end of the treatment. | 6 months after the end of the treatment.
  LV volumes (ml/m2) by Cardiac Magnetic Resonance (CMR).
Changes in LV function Changes in LV function assessed by LV volumes (ml/m2) by Cardiac Magnetic Resonance at 12 months after the end of the treatment. | 12 months after the end of the treatment.
  LV volumes (ml/m2) by Cardiac Magnetic Resonance (CMR).
Changes in LV function assessed by the presence/extent of myocardial late-enhancement at 6 months after the end of the treatment. | 6 months after the end of the treatment.
  Presence/extent of myocardial late-enhancement after gadolinium administration, in the absence of contra-indication, by Cardiac Magnetic Resonance.
Changes in LV function assessed by the presence/extent of myocardial late-enhancement at 12 months after the end of the treatment. | 12 months after the end of the treatment.
  Presence/extent of myocardial late-enhancement after gadolinium administration, in the absence of contra-indication, by Cardiac Magnetic Resonance.
Changes in LV function assessed by maximum oxygen consumption at 6 months after the end of the treatment. | 6 months after the end of the treatment.
  Maximum oxygen consumption at exercise (mL/min/kg).
Changes in LV function assessed by maximum oxygen consumption at 12 months after the end of the treatment. | 12 months after the end of the treatment.
  Maximum oxygen consumption at exercise (mL/min/kg).
Changes in LV function assessed by Natriuretic peptide plasma levels at 28 days after the end of the treatment. | 28 days after the end of the treatment.
  Natriuretic peptide plasma levels (BNP or NT-ProBNP in pg/mL).
Changes in LV function assessed by Natriuretic peptide plasma levels at 6 months after the end of the treatment. | 6 months after the end of the treatment.
  Natriuretic peptide plasma levels (BNP or NT-ProBNP in pg/mL).
Changes in LV function assessed by Natriuretic peptide plasma levels at 12 months after the end of the treatment. | 12 months after the end of the treatment.
  Natriuretic peptide plasma levels (BNP or NT-ProBNP in pg/mL).
Serious Adverse Events | 12 months
  Number of any potentially Serious Adverse Events (T-SAEs)/Reactions attributed to the experimental treatment (primary endpoint) up to 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Menasché, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital européen Georges Pompidou, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie results in publication could be shared. IPD detailed in the protocol of a planned metaanalysis could be shared
Supporting Information: Study Protocol, ICF
Time Frame: One year after the last publication
Access Criteria: Data sharing must be accepted by the sponsor and the PI based on a scientific project and scientific involvement of the PI team. Collaboration will be fostered.
  Data sharing must respect agreements made with funders. Teams wishing obtain IPD must meet the sponsor and IP team to present scientifics (and commercial) purpose, IPD needed, format of data transmission, and timeframe. Technical feasibility and financial support will be discussed before mandatory contractualization.
  Processing of shared data must comply with European General Data Protection Regulation (GDPR)

REFERENCES:
- [Background] Kervadec A, Bellamy V, El Harane N, Arakelian L, Vanneaux V, Cacciapuoti I, Nemetalla H, Perier MC, Toeg HD, Richart A, Lemitre M, Yin M, Loyer X, Larghero J, Hagege A, Ruel M, Boulanger CM, Silvestre JS, Menasche P, Renault NK. Cardiovascular progenitor-derived extracellular vesicles recapitulate the beneficial effects of their parent cells in the treatment of chronic heart failure. J Heart Lung Transplant. 2016 Jun;35(6):795-807. doi: 10.1016/j.healun.2016.01.013. Epub 2016 Jan 19. PMID 27041495
- [Background] El Harane N, Kervadec A, Bellamy V, Pidial L, Neametalla HJ, Perier MC, Lima Correa B, Thiebault L, Cagnard N, Duche A, Brunaud C, Lemitre M, Gauthier J, Bourdillon AT, Renault MP, Hovhannisyan Y, Paiva S, Colas AR, Agbulut O, Hagege A, Silvestre JS, Menasche P, Renault NKE. Acellular therapeutic approach for heart failure: in vitro production of extracellular vesicles from human cardiovascular progenitors. Eur Heart J. 2018 May 21;39(20):1835-1847. doi: 10.1093/eurheartj/ehy012. PMID 29420830
- [Background] Lima Correa B, El Harane N, Gomez I, Rachid Hocine H, Vilar J, Desgres M, Bellamy V, Keirththana K, Guillas C, Perotto M, Pidial L, Alayrac P, Tran T, Tan S, Hamada T, Charron D, Brisson A, Renault NK, Al-Daccak R, Menasche P, Silvestre JS. Extracellular vesicles from human cardiovascular progenitors trigger a reparative immune response in infarcted hearts. Cardiovasc Res. 2021 Jan 1;117(1):292-307. doi: 10.1093/cvr/cvaa028. PMID 32049348
- [Background] Lima Correa B, El Harane N, Desgres M, Perotto M, Alayrac P, Guillas C, Pidial L, Bellamy V, Baron E, Autret G, Kamaleswaran K, Pezzana C, Perier MC, Vilar J, Alberdi A, Brisson A, Renault N, Gnecchi M, Silvestre JS, Menasche P. Extracellular vesicles fail to trigger the generation of new cardiomyocytes in chronically infarcted hearts. Theranostics. 2021 Nov 2;11(20):10114-10124. doi: 10.7150/thno.62304. eCollection 2021. PMID 34815807
- [Derived] Humbert C, Cordier C, Drut I, Hamrick M, Wong J, Bellamy V, Flaire J, Bakshy K, Dingli F, Loew D, Larghero J, Fabreguettes JR, Menasche P, Renault NK, Churlaud G. GMP-Compliant Process for the Manufacturing of an Extracellular Vesicles-Enriched Secretome Product Derived From Cardiovascular Progenitor Cells Suitable for a Phase I Clinical Trial. J Extracell Vesicles. 2025 Aug;14(8):e70145. doi: 10.1002/jev2.70145. PMID 40831309